CLINICAL TRIAL: NCT01249300
Title: Comparison of Ultrasound and Videofluoroscopic Imaging Techniques in Diagnosing Dysphagia in Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Nai-Hsin Meng, China Medical University Hospital
Other Study IDs: DMR99-IRB-130
Record Dates: First submitted 2010-11-25; First posted 2010-11-29 (Estimated); Last update posted 2010-11-29 (Estimated); Status verified 2010-11

CONDITIONS: Dysphagia
Keywords: Dysphagia caused by cerebral vascular accidents
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Dysphagia: Patients with CVA which causes dysphagia
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Introduction Patients with stroke may be silent aspirators or at risk for laryngeal penetration or aspiration because of abnormal oropharyngeal functioning and thus are at risk for aspiration pneumonia and its serious effects. By providing identification of the components of the abnormal swallow, and comparing swallowing across tasks, the investigators may avoid aspiration and can instruct patients on preventative or compensatory swallowing techniques.

Materials and methods

1. Oral examination-A neurologist and speech pathologist examine the patient's swallowing function. The patient is interviewed about difficulties with food intake, chewing and swallowing during meals.
2. Ultrasound examination-Ultrasound creates image of areas inside the body using sound waves. With the patient in a sitting position, a 3/4-inch transducer (device for transmitting and receiving sound waves) is placed under the chin to visualize epiglottis movements during swallowing.
3. Modified barium swallow-While standing or sitting, the patient swallows 1/2 teaspoon of flavored barium (a radioactive substance) six times (a total of 3 teaspoons), while the tongue and pharynx (tube leading from the mouth to the esophagus) are scanned and videotaped at the same time epiglottis movement will be trace with ultrasound. The barium is given in three consistencies-thin, medium and thick (pudding-like).

The investigators will study the oral, pharyngeal and upper esophageal phases of swallow using videofluoroscopy and correlate with ultrasound tracing of epiglottis movement in patients with stroke conditions. Most of the previous studies of swallowing have utilized diagnostic imaging technique to provide a complete swallowing assessment, but limited capabilities for screening large population of patients.

INCLUSION CRITERIA: The Stroke Center inpatients and outpatients with known or suspected dysphagia can be included for study as well as patients who are admitted specifically for this protocol. (Difficulty swallowing food or pills,changed swallowing ability,coughing or choking when eating, shortness of breath during swallowing, food backing up into the mouth or nasal passage, fever or voice changes after swallowing, pain when swallowing, unexplained loss of weight.

EXCLUSION CRITERIA: Patients who are severely demented or severely compromised will be excluded if they do not have sufficient cognitive ability to follow directions. Non-ambulatory patients will be excluded if they cannot be braced or supported within the fluoroscopy unit. Highly agitated individuals will also be excluded if they are unable to remain confined in the equipment.

Analytic Methods The Student t test will be used to analyze the difference in epiglottis movements during swallowing amongst different phases. Levene's test for equality of variances will be applied to examine the variability of epiglottis movements during swallowing between the groups. All statistical analysis will be performed with SPSS.

ELIGIBILITY:
Inclusion Criteria:

* The Stroke Center inpatients and outpatients with known or suspected dysphagia can be included for study as well as patients who are admitted specifically for this protocol. (Difficulty swallowing food or pills,changed swallowing ability,coughing or choking when eating, shortness of breath during swallowing, food backing up into the mouth or nasal passage, fever or voice changes after swallowing, pain when swallowing, unexplained loss of weight.

Exclusion Criteria:

* Patients who are severely demented or severely compromised will be excluded if they do not have sufficient cognitive ability to follow directions. Non-ambulatory patients will be excluded if they cannot be braced or supported within the fluoroscopy unit. Highly agitated individuals will also be excluded if they are unable to remain confined in the equipment.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Stroke Center inpatients and outpatients with known or suspected dysphagia can be included for study as well as patients who are admitted specifically for this protocol. (Difficulty swallowing food or pills,changed swallowing ability,coughing or choking when eating, shortness of breath during swallowing, food backing up into the mouth or nasal passage, fever or voice changes after swallowing, pain when swallowing, unexplained loss of weight.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-12

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taichung, Taiwan